CLINICAL TRIAL: NCT03240367
Title: Comparison of Stapler Line Bleeding Control Techniques in Laparoscopic Gastric Bypass
Brief Title: Comparison of Stapler Line Bleeding Control Techniquessurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ersin Gündoğan (Other)
Responsible Party: Sponsor-Investigator, Ersin Gündoğan, operator doctor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/180
Record Dates: First submitted 2017-07-14; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- coutery (Experimental): Stapler bloom will be stopped with cautery
  Interventions: Other: Coutery
- clips (No Intervention): Stapler bloom will be stopped with clipping

INTERVENTIONS:
Other: Coutery — Stapler line bleeding control with coutery
  Arms: coutery

SUMMARY:
Introduction RYGB surgeon; Have become increasingly morbid obesity treatment methods with improvements in minimally invasive surgery. Ensuring patient comfort and early return to life are the criteria that should be given priority in this treatment method.The purpose of this study; Emphasizing that the cautery technique of the stapler line bleeding control methods is as successful as the other methods.

DETAILED DESCRIPTION:
The question of the availability of cautery in RYGB surgeons

ELIGIBILITY:
Inclusion Criteria:

* Morbid obese patients

Exclusion Criteria:

* Cirrhotic patients, those under 18 years of age, additional intraabdominal surgeries during LRYGBP and those who had previously undergone obesity surgery (revision surgery)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12-04 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
3-item drainage control | 8 months
  Bleeding quantities to be noted

CONTACTS AND LOCATIONS:
Overall Officials: Ersin Gündoğan, MD, Study Director — study principal investigator
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No